CLINICAL TRIAL: NCT00002445
Title: A Phase III Randomized Placebo Controlled and Double Blinded Study of IM862 for Patients With Muco-Cutaneous AIDS Associated Kaposi's Sarcoma
Brief Title: Safety and Effectiveness of an Experimental Drug, IM862, in Treating Kaposi's Sarcoma in AIDS Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cytran (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 306A; KS-20898-01; AMC-013; NCT00003879 (obsolete NCT alias)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-06

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Placebos; Sarcoma, Kaposi; Antineoplastic Agents; Treatment Outcome; Quality of Life
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; AIDS-Related Opportunistic Infections

INTERVENTIONS:
Drug: IM862

SUMMARY:
The purpose of this study is to see if it is safe and effective to use IM862 to treat Kaposi's sarcoma (KS) in AIDS patients.

DETAILED DESCRIPTION:
Patients are stratified by CD4 count, viral load, and prior systemic chemotherapy. Patients are randomized equally to receive either IM862 or placebo given intranasally every other day. Patients are seen every 4 weeks for 6 months or until disease progression to evaluate toxicity and efficacy. Quality of life is assessed before treatment, then every month for 6 months. At the end of the 6-month study evaluation period, patients with PR/CR (responders) remain on study and continue blinded treatment for an additional 6 months. For patients with stable disease (non-responders), the treatment assignment is unblinded and off-study IM862 compassionate use is offered for 6 months, regardless of treatment group. For patients with documented progressive disease (treatment failure), the treatment assignment is unblinded and off-study IM862 is offered for 6 months to any patient in the placebo group. For treatment failures in the IM862 group, IM862 is stopped and the patient is allowed other therapy options.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have AIDS-related Kaposi's sarcoma.
* Have at least 5 skin or mouth sores that do not require chemotherapy.
* Have been taking anti-HIV drugs for at least 8 weeks before study entry with no changes in the regimen.
* Are at least 18 years old.
* Agree to practice effective methods of birth control.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have an AIDS-related opportunistic infection (except for genital herpes) within 2 weeks of study entry.
* Have had another type of cancer within the past 2 years (except for certain types of skin cancer, cervical cancer, or anal cancer).
* Have a severe chest cold.
* Have certain other serious medical conditions.
* Have received certain medications, including chemotherapy, within the past 4 weeks.
* Abuse alcohol or drugs.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200

CONTACTS AND LOCATIONS:
Overall Officials: Parkash Gill, Study Chair; David Scadden, Study Chair; Ariela Noy, Study Chair
Locations (42):
- United States (31):
  - AIDS Healthcare Foundation, Los Angeles, California
  - LAGLC, Los Angeles, California
  - USC School of Medicine / Norris Cancer Hosp, Los Angeles, California
  - Tower ID Med Associates, Los Angeles, California
  - UCLA Care Ctr, Los Angeles, California
  - UCSD Med Ctr, San Diego, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Conant Med Ctr, San Francisco, California
  - Univ of Miami School of Medicine, Miami, Florida
  - BioQuan Research Group, North Miami, Florida
  - Grady Mem Hosp, Atlanta, Georgia
  - Northwestern Univ, Chicago, Illinois
  - Infectious Disease of Indiana, Indianapolis, Indiana
  - Johns Hopkins Oncology, Baltimore, Maryland
  - Massachusetts Gen Hosp, Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Med Ctr, Boston, Massachusetts
  - Washington Univ School of Medicine, St Louis, Missouri
  - UMDNJ - New Jersey Med School, Newark, New Jersey
  - St Vincents Hosp / Clinical Research Program, New York, New York
  - New York Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Columbia-Presbyterian Hosp, New York, New York
  - Albert Einstein Comprehensive Ctr, The Bronx, New York
  - Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ, Columbus, Ohio
  - Pennsylvania Oncology and Hematology Associates, Philadelphia, Pennsylvania
  - Vanderbilt Cancer Ctr, Nashville, Tennessee
  - Cytran Inc, Kirkland, Washington
  - Virginia Mason Med Ctr, Seattle, Washington
  - Univ of Washington / Harborview Med Ctr, Seattle, Washington
- Australia (4):
  - St Vincent's Hosp / Dept of Haematology, Darlinghurst
  - Alfred Hosp, Prahan
  - Prince of Wales Hosp, Randwick
  - Taylors Square Clinic, Sydney
- Belgium (2):
  - Inst of Tropical Medicine, Antwerp
  - CHU Saint Pierre, Brussels
- Canada (5):
  - BC Cancer Agency, Vancouver, British Columbia
  - Ottawa General Hospital, Ottawa, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Toronto Gen Hosp, Toronto, Ontario
  - Montreal Gen Hosp / Div of Clin Immuno and Allergy, Montreal, Quebec